CLINICAL TRIAL: NCT01625013
Title: Long-Term Management of "Younger, Active" Patients With Pain From Early Knee Osteoarthritis With Synvisc-One (Hylan G-F 20)
Brief Title: Synvisc-One for Younger, Active Patients With Osteoarthritis
Acronym: SYNVISC-ONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anthony Luke (Other)
Responsible Party: Sponsor-Investigator, Anthony Luke, Associate Professor of Clinical Orthopaedic Surgery, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSF-SYNVISC-ONE 001
Record Dates: First submitted 2012-06-11; First posted 2012-06-21 (Estimated); Results first posted 2020-03-27 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-04

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; viscosupplementation; Active; Knee; Synvisc-One
MeSH Terms: conditions — Osteoarthritis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Synvisc-One (Experimental)
  Interventions: Device: Synvisc-One (G-F 20)

INTERVENTIONS:
Device: Synvisc-One (G-F 20) — Synvisc G-F 20 will be injected in the symptomatic knee using a standard supine lateral approach using a 20-gauge needle. Patients will be treated at baseline and followed out to three years. Patients may return for retreatment as early as 4 months post their prior injection if they meet the retreatment criteria pain levels for Worst Knee Pain. If the subjects need another injection, the follow-up cycle will restart at Visit 1 and the subject will be seen every 6 months and followed-up for 3 years.

SUMMARY:
This study aims to study use of viscosupplementation as a treatment of pain for young individuals who are active. Typically viscosupplementation is considered an intervention for knee osteoarthritis often for older patients who are less active. Many young active patients can also develop knee osteoarthritis after trauma or surgery or for congenital reasons. Treatment of these patients commonly are steroid injections which have more biologically detrimental effects for cartilage compared to viscosupplementation Synvisc One injections which are a single injection will be used to determine effectiveness of reducing pain and maintaining an active healthy lifestyle for younger patients aged 30-50 years old.

DETAILED DESCRIPTION:
This study will be an open label longitudinal cohort study with natural history over 3 years. Screening data will be reviewed to determine subject eligibility. Subjects who meet all inclusion criteria and none of the exclusion criteria will be entered into the study. Subjects enrolled in the cohort will have baseline functional testing performed including a motion gait analysis, 12 minute walk test, and 3-day accelerometer data. Subjects will receive a single 6 mL intra-articular injection of hylan G-F 20 in the target knee at baseline. All ongoing treatments will be monitored at 6 month intervals over the 3 year duration of the study. Patients can receive any other conservative treatments (e.g., oral medications, physical or other therapy, acupuncture, etc., except other injection treatments) and current treatments will be documented during each patient encounter. An initial injection of hylan G-F 20 will be injected in the symptomatic knee using a standard supine lateral approach using a 20 gauge needle. A face to face follow up visit will be carried out 6 months after first injection with additional face to face meetings every 6 months thereafter unless the subject requires an additional injection of hylan G-F 20. Hylan G-F 20 treatments can be administered up to three times each year during the study duration. After each injection, follow up measures will be carried out using secure e-mail or phone contact at 6 weeks, 12 weeks, 18 weeks after each in-office evaluation or injection. Follow up will consist of WOMAC, Lysholm score, and Tegner score. Patients may return for retreatment of hylan G-F 20 if symptoms recur after at least 4 months following their previous injection and they meet the inclusion criteria with pain levels of WOMAC A1, C8, C9, C10 and/or C23 equaling 2 or more. Patients requiring three injections of hylan G-F 20 in 4 months or less will be allowed to exit the cohort after their six-month follow up following the third injection. Otherwise, patients will be followed until they reach the 3 year follow up, or drop out for other injection treatments or surgical treatment. Therefore, patients would potentially be able to receive up to 9 injections during the 3 year study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 30-50 years
* History of symptomatic unilateral primary or secondary knee OA for more than 6 months
* Signed written informed consent
* Radiographic evidence of Kellgren-Lawrence Grade I or II OA of the target knee
* Body Mass Index (BMI) < 30 kg/m2
* Activity criteria (Tegner score > 3)
* Continued target knee OA pain despite conservative treatment ≥ 3 months (e.g., weight reduction, physical therapy, analgesics)
* Willing to withhold intake of NSAIDs (including COX-2 inhibitors) and analgesics, for a washout period of minimum 3 days up to 21 days prior to baseline visit (depending on medication)
* Willing to discontinue prohibited treatments and medications throughout study period

Baseline inclusion criteria

* Completed OA medication washout period
* Target knee pain 4-8 (0-10 NRS) during most painful knee movement (Worst Knee Pain)
* If female, must have had a negative urine pregnancy test and used a medically acceptable form of contraception for at least 1 month prior to baseline and agree to continued use of contraception for the duration of the study. Otherwise, females must be surgically sterile, or postmenopausal (as documented in medical history) for at least 1 year. The fetal safety profile for G-F 20 is unknown. Pregnancy will affect the individual's regular activity levels. Females who become pregnant during the study will be excluded from the study. Subjects who become pregnant will be followed up by telephone every 3 months to check for any adverse effects. They will also be recommended to follow routine obstetric visits. Males should be able to father children as it has no expected effects on activity levels.

Exclusion Criteria:

* Known allergy to hylan G-F 20 or any of its components, or to avian proteins, eggs, feathers, down, or poultry
* Clinically apparent tense effusion or other acute inflammation of the target knee at baseline
* History of target knee viscosupplementation treatment
* History of major surgery for OA in target knee including arthroplasty or tibial osteotomy
* Arthroscopic surgery or intraarticular steroid injection in target knee within six months of baseline visit
* Significant (as judged by the Investigator) alignment deformity of target knee
* Ipsilateral symptomatic OA of hip or ankle; contralateral symptomatic OA of hip, knee, or ankle

History of:

* Septic OA of any joint
* Inflammatory arthropathy such as RA, gout, pseudogout, lupus, crystalline inflammatory arthropathy
* Active infection of lower extremity
* Known significant acute and/or concurrent medical disease including, but not limited to current malignancy, history of transplant surgery, congestive heart failure, significant unstable cardiovascular disease, renal hepatic pulmonary, endocrine, metabolic, or GI condition
* Any known contraindication to acetaminophen
* Venous or lymphatic stasis in either leg
* Peripheral vascular disease
* Patient has been prescribed chronic opioid analgesics at time of baseline visit
* Concurrent multi-system or multi-limb trauma
* Patient plans to become pregnant during study period
* Patient plans to move significantly out of area, have surgery, or initiate or cease other OA treatments
* Knee pain improves during washout period
* Workman's Comp patient

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2017-10-02 (Actual); Study Completion 2019-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Luke, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Synvisc-One
Started | 51
Completed | 48
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Synvisc-One
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 32
  More than one race | 0
  Unknown or Not Reported | 11

OUTCOME MEASURES:

1. Primary Outcome: "Worst Knee Pain" Likert Scale (0-10) Reported on Survey
Description: Worst Knee Pain Scores were measured using a "Worst Knee Pain" Likert scale, the score ranges from 0-10, zero indicating no pain and 10 indicating the worst pain.
  Patient Acceptable Symptom State (PASS) is a "Worst Knee Pain" reported score of less than 4 to be "positive". Patient Acceptable Symptom State (PASS) is the highest level of symptom beyond which patients consider themselves well.
  Minimum Clinical Important Improvement (MCII) is improvement at any time in the 26 week time frame that "Worst Knee Pain" is reported at 2 points less than baseline.
Time Frame: 26 weeks after injection at baseline
Population: Patients at 26 weeks post-injection Number 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synvisc-One
Number analyzed (Participants) | 43
Participants
  Patient Acceptable Symptom State (PASS) | 25
  Minimum Clinical Important Improvement (MCII) | 35

2. Secondary Outcome: Patient Acceptable Symptom Score (The Effect of Repeated Treatments)
Description: Though symptoms can be improved for periods up to 6 months, pain symptoms can recur. The effect of repeated treatments of hylan G-F 20 will be studied with the Patient Acceptable Symptom Score less than 4/10 for the reported Worst Knee Pain score on follow up surveys.
  Worst Knee Pain Scores were measured using a "Worst Knee Pain" Likert scale, the score ranges from 0-10, zero indicating no pain and 10 indicating the worst pain.
  Patient Acceptable Symptom State (PASS) is a "Worst Knee Pain" reported score of less than 4 to be "positive". Patient Acceptable Symptom State (PASS) is the highest level of symptom beyond which patients consider themselves well.
Time Frame: 26 weeks post-injection Number 2, an average of 52 weeks
Population: Patients receiving Synvisc One injection Number 2
Measure: Count of Participants; unit: Participants
Groups:
- Synvisc-One Second Injection: Synvisc-One (G-F 20): Synvisc G-F 20 will be injected a second time in the symptomatic knee using a standard supine lateral approach using a 20-gauge needle. Patients will be treated at baseline and followed out until three years from their first injection. Patients may return for retreatment as early as 4 months post their prior injection if they meet the retreatment criteria pain levels for Worst Knee Pain. If the subjects need another injection, the follow-up cycle will restart at Visit 1 and the subject will be seen every 6 months and followed-up for a total of 3 years.
Arm/Group | Synvisc-One Second Injection
Number analyzed (Participants) | 37
Participants
  Patient Acceptable Symptom State < 4/10 worst knee pain | 0
  Patient Acceptable Symptom State > 4/10 | 18
  Missing Data | 19

3. Secondary Outcome: Minimal Clinical Important Improvement (The Effect of Repeated Injections)
Description: Though symptoms can be improved for periods up to 6 months, pain symptoms can recur. The effect of repeated treatments of hylan G-F 20 will be studied with the Minimal Clinical Important Improvement less than 2 points from baseline on a 10-point likert scale for the reported Worst Knee Pain score on any follow up survey within 3 months. Worst Knee Pain Scores were measured using a "Worst Knee Pain" Likert scale, the score ranges from 0-10, zero indicating no pain and 10 indicating the worst pain. Patients can reinject after 4 months.
Time Frame: up to 15 months (within 3 months from the second Synvisc One injection)
Population: Patients receiving Synvisc One injection Number 2
Measure: Count of Participants; unit: Participants
Arm/Group | Synvisc-One Second Injection
Number analyzed (Participants) | 37
Participants
  Minimal Clinical Important Improvement more than 2 points improvement from baseline | 10
  MCII less than 2 points improvement from baseline | 12
  Missing Data | 15

4. Secondary Outcome: Identify the Effects of Treatment on Activity Levels
Description: To identify the effects of treatment with hylan G-F 20 on activity levels (using objective activity measures utilizing accelerometer and Physical Activity Enjoyment Scale (PACES) and quality of life scores (WOMAC, SF-12) comparing baseline to treatment at 3 months.
Time Frame: 26 weeks post-injection at baseline through 3 years post-injection
Population: The minimal data collected are invalid due to end user error and inaccurate data collection practices, therefore no valid data exist to report.
Arm/Group | Synvisc-One Second Injection
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at 6, 12, and 18 weeks after each injection/clinic visit, up to 3 years for each participant.
Arm/Group | Synvisc-One
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 29/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Synvisc-One (N=51)
Severe Swelling, Pain, and/or Stiffness (Musculoskeletal and connective tissue disorders) | 27
Reinjury (Musculoskeletal and connective tissue disorders) | 2 — 1 knee reinjury while playing sports; 1 reinjury while twisting knee, leading to meniscus tear

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-05-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT01625013/Prot_SAP_001.pdf